CLINICAL TRIAL: NCT04538391
Title: Bupivacaine Versus Meloxicam Infiltration on Post Cesarean Section Pain Relief
Brief Title: Intra Incisional Infiltration of Bupivacaine Versus Meloxicam on Post Cesarean Section Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, Lecturer of obstetrics and gynecology, Menoufia Obstetrics and Gynecology Group
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12/2019OBSGN38
Record Dates: First submitted 2020-08-24; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section Pain

STUDY DESIGN:
Intervention Model Description: Group A (bupivacaine group): included 35 patients in which and subcutaneous tissue (upper and lower flaps) were infiltrated with 20 ml of 0.25% bupivacaine hydrochloride. (Marcaine, 25% vial, Astra Zeneca) diluted in 20 ml of 0.9% saline.
  Group B (meloxicam group): included 35 patients in which and subcutaneous tissue (upper and lower flaps) were infiltrated with meloxicam 15mg (Anticox 2 ampoule 15mg/3ml, ADWIA Pharmaceuticals). diluted in 20 ml of 0.9% saline.
  Group C (placebo group): included 35 patients in which skin and subcutaneous tissue was infiltrated with 20 ml 0.9% saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each woman received a disposable syringe containing a medication corresponding to her order of participation in the trial. Packing. Sealing and numbering were performed by health care provider who did not actively share in the process of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bupivacaine group (Active Comparator): included 35 patients in which and subcutaneous tissue (upper and lower flaps) were infiltrated with 20 ml of 0.25% bupivacaine hydrochloride. (Marcaine, 25% vial, Astra Zeneca) diluted in 20 ml of 0.9% saline.
  Interventions: Drug: local ifiltration Bupivacaine, Meloxican and placebo
- meloxicam group (Active Comparator): included 35 patients in which and subcutaneous tissue (upper and lower flaps) were infiltrated with meloxicam 15mg (Anticox 2 ampoule 15mg/3ml, ADWIA Pharmaceuticals). diluted in 20 ml of 0.9% saline.
  Interventions: Drug: local ifiltration Bupivacaine, Meloxican and placebo
- placebo group (Active Comparator): included 35 patients in which skin and subcutaneous tissue was infiltrated with 20 ml 0.9% saline.
  Interventions: Drug: local ifiltration Bupivacaine, Meloxican and placebo

INTERVENTIONS:
Drug: local ifiltration Bupivacaine, Meloxican and placebo — no other intervention done

SUMMARY:
Investigation: compare the effect of local infiltration of incision site with bupivacaine and local infiltration with meloxicam in women undergoing cesarean sections on postoperative pain relief and analgesic requirement.

Condition: post cesarean sections analgesia intervention: infiltration of incision bupivacaine versus meloxicam Phase: Not applicable

DETAILED DESCRIPTION:
study type: randomized clinical trial actual enrollment: 119 allocation: Random intervention model: three groups assignment masking: open lebal primary purpose: pain relief after Cesarean section actual study start: March 3, 2019 Primary Completion: March 5, 2020 actual study completion date: May 9, 2020

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-40 years
* Elective C.S at term
* Patient having no medical disorders
* Patient with no obstetrical complications

Exclusion Criteria:

* extreme of reproductive age
* allergy to local anesthetic infiltration agent
* any medical disorders or obstetrical complications as ante partum hemorrhag, pre-eclampsia
* refusal to participate in the trial.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | immediately after the intervention
  Assessment of pain scores after Cesarean section
Postoperative analgesic requirements | immediately after the intervention
  Assessment of Postoperative analgesic requirements
time of first dose of analgesia | immediately after the intervention
  Determination of time of first dose of analgesia

SECONDARY OUTCOMES:
Postoperative fever | immediately after the intervention
  Assessment of Postoperative fever
onset of mobilization | immediately after the intervention
  Assessment of onset of mobilization
side effects of medications | immediately after the intervention
  Assessment of side effects of medications
Pain assessment by visual analogue scale | immediately after the intervention
  Post-operative pain assessment was done using a 10-point visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Anter, MD, Principal Investigator — Menoufia University hospital
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
through the E-maill address